CLINICAL TRIAL: NCT01667172
Title: Study of Technical Accuracy and Userfriendliness of Two Point-of-care C Reactive Protein Devices
Brief Title: Technical Accuracy and Userfriendliness of Two Point-of-care C Reactive Protein Devices in Comparison With Laboratory CRP Testing.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Jan Verbakel, Research Assistant, KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: S54271
Record Dates: First submitted 2012-08-14; First posted 2012-08-17 (Estimated); Last update posted 2012-08-17 (Estimated); Status verified 2012-08

CONDITIONS: Healthy and Acutely Ill Children & Adults

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (1):
- point-of-care test for CRP (Other)
  Interventions: Device: Point-of-Care C Reactive Protein measurement on capillary blood

INTERVENTIONS:
Device: Point-of-Care C Reactive Protein measurement on capillary blood — capillary blood fingerstick method to determine C Reactive Protein level in the blood

SUMMARY:
Study to test technical accuracy and userfriendliness of two Point-of-care C Reactive Protein devices (POC CRP devices) in comparison with laboratory CRP testing on children and adults.

Research questions:

1. Are the POC CRP devices technically accurate? Do the measured values agree with CRP values measured at the clinical laboratory?
2. Are the 2 POC CRP devices equivalent ? 2.1. Are the 2 POC CRP devices equally reliable? 2.1.1. Comparison of 2 measurements in the same patient on 1 device (inter-observer-variability) 2.1.2. Comparison of 2 measurements in the same patient on 2 identical devices (inter-device-variability) 2.2. Are the 2 Point-of-Care CRP devices equally userfriendly in a general practice surgery? (userfriendliness

ELIGIBILITY:
Inclusion Criteria:

* children: aged 1 month to 14 years
* adults: aged 18-65 years

Exclusion Criteria:

* children and adults not understanding Dutch language

Ages: 1 Month to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2012-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
technical accuracy | 3 months
  correlation obtained between the results from the Point-of-care C Reactive Protein devices and the results from the laboratory

SECONDARY OUTCOMES:
User-friendliness | 3 months
  evaluation of the userfriendliness by General Practitioners at 5 practices, on a five point Likert-scale scoring these criteria: device start-up, test duration, sample size, test characteristics, calibration, measuring range, handling of test tubes, filling of the capillary, placing the test cartridge, test recording and additional material usage. The median results are compared between both devices qualitatively.
Inter-device variability | 3 months
  The inter-device-variability (by 1 physician) was tested on 10 patients in one General Practice surgery each on two different Point-of-Care devices of the same brand.
Inter-observer variability | 3 months
  The inter-observer variability (by two physicians) was tested on 10 patients in one GP surgery on two different Point-of-care devices of the same brand.

CONTACTS AND LOCATIONS:
Locations (3):
- Belgium (3):
  - Huisartspraktijken, Leuven, Vlaams-Brabant
  - Medisch Centrum voor Huisartsen, Leuven, Vlaams-Brabant
  - UZ Leuven, Leuven, Vlaams-Brabant

REFERENCES:
- [Background] Van den Bruel A, Thompson MJ, Haj-Hassan T, Stevens R, Moll H, Lakhanpaul M, Mant D. Diagnostic value of laboratory tests in identifying serious infections in febrile children: systematic review. BMJ. 2011 Jun 8;342:d3082. doi: 10.1136/bmj.d3082. PMID 21653621
- [Background] Van den Bruel A, Haj-Hassan T, Thompson M, Buntinx F, Mant D; European Research Network on Recognising Serious Infection investigators. Diagnostic value of clinical features at presentation to identify serious infection in children in developed countries: a systematic review. Lancet. 2010 Mar 6;375(9717):834-45. doi: 10.1016/S0140-6736(09)62000-6. Epub 2010 Feb 2. PMID 20132979